CLINICAL TRIAL: NCT04474223
Title: Surveillance and Treatment to Prevent Fetal Atrioventricular Block Likely to Occur Quickly (STOP BLOQ)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-00363
Record Dates: First submitted 2020-07-14; First posted 2020-07-16 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: AVB - Atrioventricular Block; Fetal AVB
MeSH Terms: conditions — Atrioventricular Block | interventions — Dexamethasone; Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mothers with Fetuses Who Have 2° AVB or AV interval > 170ms (Experimental)
  Interventions: Drug: Dexamethasone; Drug: IVIG

INTERVENTIONS:
Drug: Dexamethasone — In mother in whom 2° AVB or AV interval >170 ms has been diagnosed in the fetus:
  Dexamethasone 8 mg po/day for 10 days. Then dexamethasone 4 mg po/ day through 28 weeks 6 days gestational age (GA); then 3 mg/day from 29 wks 0 days to 29 wks 6 days GA; then 2 mg/day until delivery
Drug: IVIG — In a mother in whom 2° AVB has been diagnosed in the fetus:
  One dose of IVIG [1g/kg of maternal weight (max dose 70 g)] at diagnosis of 2° AVB (within 12 hours of detection by mother via home monitoring and within 6 hours of confirmation by echocardiogram). A fetal AV interval > 170 ms will not be treated with maternal IVIG, only dexamethasone.

SUMMARY:
Fetal complete (i.e., third degree, 3°) atrioventricular block (AVB), identified in the 2nd trimester of pregnancy in an otherwise normally developing heart, is almost universally associated with maternal anti-Ro autoantibodies and results in death in a fifth of cases. To date treatment of 3° AVB has been ineffective in restoring normal rhythm (NR) which may be because current surveillance is limited to once- weekly fetal echocardiograms. It is hypothesized that there may be a vital transition period of several hours in which incomplete block (2° AVB) may be successfully treated avoiding fully advanced irreversible 3° AVB. To optimize the likelihood of timely detection of the transition period this study comprises three steps: 1) to risk stratify for high titer anti-Ro antibodies, which are necessary but not sufficient to develop fetal AVB; 2) to empower mothers to identify 2° AVB by using fetal heart rate and rhythm monitoring (FHRM) at home, and 3) to rapidly treat mothers who detect an abnormality by monitoring with an urgent echocardiogram that confirms 2° AVB with the hope of reversing 2° AVB before it becomes permanent (3° AVB). In addition, it will be determined if FHRM reduces the need for weekly echoes. Although mothers with low titer anti-Ro will not be continued in Step 2 and therefore not followed by FHRM, birth ECGs will be collected to confirm that low titer antibodies do not confer risk. It is anticipated that this study will provide an evidenced based surveillance strategy for those mothers at high risk of having a child with 3° AVB.

DETAILED DESCRIPTION:
Fetal complete (3°) atrioventricular block (AVB), identified in the 2nd trimester in an otherwise normally developing heart, is almost universally associated with maternal anti-Ro autoantibodies, which transcytose the placenta via the trophoblastic IgG receptor, FcγRn. The burden of 3° AVB is considerable: perinatal mortality of 18% exceeds that for all non-cardiac congenital anomalies combined, and almost all survivors require lifelong cardiac pacing with its associated complications. It has been speculated that full expression of conduction disease occurs by sequential fetal progression from normal rhythm (NR) to 1° AVB [prolonged AV interval assessed by echocardiogram (echo)], to 2° AVB (irregular cardiac rhythm or bradycardia), culminating in 3° AVB. Fetal heart rate and rhythm monitoring (FHRM) suggests a time interval of ~12 hours for the transition from NR to 3° AVB, albeit the culprit biologic processes (inflammation leading to fibrosis) likely initiate prior to clinical detection. Anecdotal evidence suggests this transition period, marked by an irregular rhythm and/or bradycardia, may be the only window of opportunity for anti-inflammatory treatment to restore NR.

A barrier to preventing progression to 3° AVB is the absence of a technique to accurately surveil for the precipitate transition from NR to 3° AVB. Surveillance limited to weekly echos (current standard of care) may be too infrequent to detect this transition period when treatment is most likely to be effective. We have now obviated this obstacle and shown that ambulatory FHRM by the mother at home with confirmation of abnormal findings by echo is not only feasible but may afford rapid treatment restoring NR. Combining results from studies comprising 275 anti-Ro+ pregnancies, 87% completed monitoring with a false positive rate of 5%. In 4 cases of 2° AVB identified by FHRM and treated <12h, AVB reversed. Remarkably, no cases of 2° or 3° AVB were missed, suggesting mothers can recognize abnormal FHRM, reducing or precluding the need for weekly echos.

The proposed project combines the expertise of fetal cardiologist Bettina F. Cuneo, MD, initiator and PI of the FHRM program, and rheumatologist Jill P. Buyon, MD, founder/director of the largest extant registry of anti-Ro-mediated AVB, whose research on the pathogenesis supports a fetal inflammatory component associated with high-titer antibodies. Participants will be referred from 35 sites in 3 sequential Steps: 1) Screening for high titer anti-Ro60 or Ro52 centrally in Dr. Buyon's lab; 2) Surveillance by FHRM 3x daily and weekly echo; 3) Treatment of 2° AVB identified by FHRM confirmed by echo. Feasibility of FHRM supported by weekly echo of high-autoantibody-titer mothers will be leveraged to address the efficacy of expeditious (<12 h after detection) treatment of 2° AVB as well as the incidence/outcome of AV interval prolongation and extra-nodal disease.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Be <18 weeks pregnant at the time of enrollment
4. Titer of anti-Ro 52 or 60 antibodies ≥1,000 EU
5. Any positive titer of anti-Ro if a history of a previously affected child
6. Ability to take oral medication and be willing to adhere to the dexamethasone and IVIG protocols.
7. Ability to perform Doppler fetal heart rate and rhythm monitoring in the ambulatory setting,
8. Ability to send an audiotext message by cell phone therefore the participant will be informed that they need a phone with texting capabilities. Located within 6 hours drive of the participating pediatric cardiology site
9. Be ≥18 years of age

Exclusion Criteria:

1. Multi-fetal pregnancy
2. Known allergic reactions to components of IVIG, or dexamethasone or maternal IgA deficiency
3. Fetal conduction system disease already present in the current pregnancy
4. Any women who in the opinion of the investigator cannot understand the consent form or be able to perform thrice daily home monitoring or recognize an abnormal fetal heart rate or rhythm
5. Women prisoners
6. Treatment with >20 mg/prednisone q day or with any dose of fluorinated steroids at enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Must be <18 weeks pregnant at the time of enrollment
Enrollment: 1300 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of 2° AVB subjects with NR (1:1 AV conduction) at birth | up to 25 weeks post-enrollment
  The presence of NR (normal rhythm) will be determined by electrocardiogram (ECG)

SECONDARY OUTCOMES:
Percentage of 2° AVB subjects who maintain NR at age 1 year. | 1 year post-birth
  The presence of NR will be determined by ECG
Percentage of AV interval > 170 msec subjects with NR at birth | At birth
  AV intervals will be determined by EKG
Incidences of isolated extra-nodal cardiac disease | up to 1 year post-birth
  Extra-nodal cardiac disease includes: Endocardial fibroelastosis, dilated cardiomyopathy, and AV valve insufficiency. Isolated exta-nodal cardiac disease will be determined by echocardiogram.

CONTACTS AND LOCATIONS:
Overall Officials: Jill Buyon, MD, Principal Investigator — NYU Langone Health; Bettina Cuneo, MD, Principal Investigator — University of Colorado, Denver
Locations (24):
- United States (23):
  - Phoenix Children's Hospital/Dignity Health, Phoenix, Arizona
  - University of California - Los Angeles (UCLA), Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of California-San Francisco, San Francisco, California
  - University of Colorado, Denver (UCD), Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Children's National Medical Center/George Washington University, Washington D.C., District of Columbia
  - University of Kentucky / Kentucky Children's Hospital, Lexington, Kentucky
  - University of Louisville / Norton Children's Hospital, Louisville, Kentucky
  - University of Michigan / C. S. Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Minnesota, Minneapolis, Minnesota
  - Perinatal Associates of New Mexico, Rio Rancho, New Mexico
  - NYU Langone Health, New York, New York
  - Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - UH Rainbow Babies / Children's Hospital, Cleveland, Ohio
  - Cleveland Clinic Lerner College of Medicine, Cleveland, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - University of Utah Health, Salt Lake City, Utah
  - University of Vermont Children's Hospital, Burlington, Vermont
  - Eastern Virginia Medical School (EVMS), Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
- Stollery Children's Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposes to use the data will have access to the data upon reasonable request and when a stated purpose and approval by a committee is provided. Requests should be directed to Jill.Buyon@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.